CLINICAL TRIAL: NCT04482816
Title: Randomized Study of Physiological vs Right Ventricular Pacing in Patients With Normal Ventricular Function Post-TAVI (PHYS-TAVI Trial)
Brief Title: Physiological vs Right Ventricular Pacing in Patients With Normal Ventricular Function Post-TAVI
Acronym: PHYS-TAVI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Josep Lluis Mont Girbau (Other)
Responsible Party: Sponsor-Investigator, Josep Lluis Mont Girbau, Head of Arrhythmia Section. Professor of Cardiology, Hospital Clinic of Barcelona
Organization: Hospital Clinic of Barcelona (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PHYS-TAVI TRIAL
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-12

CONDITIONS: Transcatheter Aortic Valve Implantation; Physiological Pacing; Right Ventricular Pacing; AV Block
Keywords: TAVI; Physiological Pacing; AV Block
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be explained to be randomized to either of the two branches. The type of therapy applied will not be communicated to the patient. The follow-up will be the same in the two branches. During the visits, it will not be said which therapy has been applied.
  The echocardiographer and the follow-up by the Hemodynamic Team will be blind.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physiological pacing (Experimental): Lead placed in the His-Purkinje system (his or branch) in order to achieve QRS shortening and physiologic pacing. A backup lead will be implanted in the right ventricle.
  If hisian pacing is not achieved (QRS is not shortened > 20% or QRS is not <130ms), the left bundle branch will be paced according to the criteria established in the literature (right branch block and intrinsic deflection <85ms).
  Crossover from physiological pacing to right ventricular pacing will be allowed in the following situations: failed physiological pacing lead implantation; high thresholds (>3.5V / 1ms); no shortening of QRS (shortening <20%) or failure to meet non-selective HBP criteria or left bundle branch pacing criteria.
  Interventions: Device: Physiological pacing
- Right ventricular pacing (Active Comparator): Lead placed in the right ventricle (conventional pacing).
  Interventions: Device: Right ventricular pacing

INTERVENTIONS:
Device: Physiological pacing — Pacing of the his bundle or the left bundle branch
  Arms: Physiological pacing
Device: Right ventricular pacing — Conventional pacing; right ventricular pacing
  Arms: Right ventricular pacing

SUMMARY:
Single-center randomized trial in patients with pacing indication (AV block) after TAVI (transfemoral aortic valve implantation) and LVEF> 50%, that aims to study the percentage of patients who improve at 12 months in a combined clinical endpoint.

DETAILED DESCRIPTION:
There is currently no evidence of the best mode of definitive pacing after TAVI in patients with preserved systolic ventricular function and AV block. Through this study, investigators intend to elucidate the best post TAVI pacing strategy, comparing the effect of right apical pacing vs. physiological pacing on the evolution of both echocardiographic and clinical parameters.

Investigators will include 24 patients without ventricular dysfunction (LVEF> 50%) and with AV block pacing indication after TAVI.

Patients will be randomized to 2 types of pacing (parallel randomized trial): physiological or right ventricular pacing (conventional).

PHYS-TAVI trial will analyze the following parameters in the 2 groups: survival; NYHA class; distance in the 6-minute walking test; hospital admissions; left ventricular function; echocardiographic asynchrony (strain and flash septal); NTproBNP; and quality of life/symptoms with the Kansas City Cardiomyopathy Questionnaire test (KCCQ-12)

Clinical, and echocardiographic follow-up will be performed for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Successful implantation of TAVI according to VARC-2 criteria.
* Indication of cardiac pacing due to AV block according to ESC Guidelines.
* LVEF> 50%.
* The patient must indicate their acceptance to participate in the study by signing an informed consent document.

Exclusion Criteria:

* Ventricular dysfunction: LVEF <50%.
* Transapical TAVI.
* Participating currently in a clinical investigation that includes an active treatment.
* Patients with left bundle branch block but without indication of pacing (AV block).
* Life expectancy <12 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Clinical combined endpoint: survival; and improvement > 1 point in NYHA class or > 25% increase in the distance covered in the 6-minute walking test. | 12 months
  Determine the percentage of patients who improve at 12 months on a clinical combined endpoint: survival; and improvement > 1 point in NYHA class or > 25% increase in the distance covered in the 6-minute walking test.

SECONDARY OUTCOMES:
Change in left ventricular ejection fraction. | 12 months
  Left ventricular ejection fraction (LVEF %) measured with Simpson method with echocardiography (Delta left ventricular ejection fraction: 12 months LVEF - baseline LVEF).
Correction of echocardiographic asynchrony: septal flash expressed in mm. | 30 days; 12 months
  Correction of septal flash determined with echocardiography (M mode).
Distance covered in the 6-minute walking test. | 30 days; 12 months
  Distance in meters walked in 6 minutes.
Change in NYHA functional class. | 30 days; 12 months
  NYHA functional class I, II, III, IV.
Change in degree of mitral regurgitation. | 12 months
  Mitral regurgitation measured with echocardiography.
Change in NTproBNP. | 30 days; 12 months
  NTproBNP blood levels.
Hospitalization due to heart failure. | 12 months
  Hospitalization: patient hospitalization (yes/no).
QRS duration | Implant; 12 months
  QRS duration (milliseconds) measured with a 12-lead ECG (in the electrophysiology lab polygraph)
Score on quality of life/symptoms Questionnaire (KCCQ-12 Kansas City Cardiomyopathy Questionnaire ) | 30 days; 12 months
  Score in KCCQ-12: higher=better.
Correction of global longitudinal strain | 30 days; 12 months
  Global longitudinal strain assessed with two-dimensional speckle-tracking echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: José M Tolosana, MD, PhD, Principal Investigator — Institut Clínic Cardiovascular (ICCV), Hospital Clínic Barcelona.; Margarida Pujol Lopez, MD, Principal Investigator — Institut Clínic Cardiovascular (ICCV), Hospital Clínic Barcelona.; Lluís Mont, MD, PhD, Study Director — Institut Clínic Cardiovascular (ICCV), Hospital Clínic Barcelona.; Eduard Guasch, MD, PhD, Study Chair — Institut Clínic Cardiovascular (ICCV), Hospital Clínic Barcelona.
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pujol-Lopez M, Regueiro A, Graterol FR, Garcia-Ribas C, Uribe L, Jimenez-Arjona R, Borras R, Guasch E, Guichard JB, Carballeira L, Falzone PV, Regany-Closa M, Casal R, Poza M, Arbelo E, Porta-Sanchez A, Roca-Luque I, Sitges M, Doltra A, Tolosana JM, Mont L. Left Bundle Branch Versus Apical Pacing in Atrioventricular Block and Normal Cardiac Function Post-transcatheter Aortic Valve Implantation: PhysTAVI Trial. CJC Open. 2025 Jul 30;7(12):1610-1620. doi: 10.1016/j.cjco.2025.07.014. eCollection 2025 Dec. PMID 41542133